CLINICAL TRIAL: NCT03759821
Title: Engaging Fathers for Effective Child Nutrition and Development in Tanzania (EFFECTS): A Community-Based Bundled Nutrition and Parenting Intervention
Brief Title: Engaging Fathers for Effective Child Nutrition and Development in Tanzania
Acronym: EFFECTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Project Concern International (Other)
Collaborators: Purdue University (Other); Harvard School of Public Health (HSPH) (Other); Africa Academy for Public Health (Other); The Eleanor Crook Foundation (Unknown); Conrad N. Hilton Foundation (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Principal Investigator, Mary Pat Kieffer, Senior Director for Health, Project Concern International
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 01
Record Dates: First submitted 2018-10-27; First posted 2018-11-30 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Child Nutrition and Early Child Development
Keywords: Infant and young child feeding; Nutrition; Stimulation; Parenting; Early childhood development; Social and behavior change; Father involvement; Male engagement; Household decision-making; Community health workers; Peer groups; Integrated interventions
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Eighty villages in the Mara region of Tanzania will be randomly selected and randomly allocated with equal probability and in equal numbers to one of the five EFFECTS study arms. In each participating village, one sub village will be randomly selected with equal probability, and a sampling frame of all households in that sub village will be created with the help of local leaders. Households will be selected from this sampling frame using simple random sampling. The selected households will be listed in random order and visited by study staff, who will assess whether a household meets all inclusion criteria and provides informed consent. Households will be visited until 12 households are enrolled in each village. If not enough eligible households are found, additional households will be selected using the same procedure from the nearest sub village in the same village.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Nutrition, mothers (Experimental): Community health workers (CHWs) will facilitate peer group sessions with mothers of children aged 0-18 months at enrollment. The CHWs will deliver key messages and facilitate problem-solving and skill-building activities to promote nutrition-related behavior change. Group sessions will last between 1.5-2 hours and groups will meet biweekly for a period of 12 months. Due to the COVID pandemic, group sessions were paused for three months (March-June 2020). The intervention resumed in July 2020 with delivery via home visits rather than peer groups, and concluded in September 2020.
  Interventions: Behavioral: Nutrition, mothers
- Nutrition, mothers and fathers (Experimental): Community health workers (CHWs) will facilitate peer group sessions with mothers and fathers of children aged 0-18 months at enrollment. The CHWs will deliver key messages and facilitate problem-solving and skill-building activities to promote nutrition-related behavior change. Group sessions will last between 1.5-2 hours and the groups will meet biweekly for a period of 12 months. Due to the COVID pandemic, group sessions were paused for three months (March-June 2020). The intervention resumed in July 2020 with delivery via home visits rather than peer groups, and concluded in September 2020.
  Interventions: Behavioral: Nutrition, mothers and fathers
- Nutrition+parenting, mothers (Experimental): Community health workers (CHWs) will facilitate peer group sessions with mothers of children aged 0-18 months at enrollment. CHWs will deliver key messages and facilitate problem-solving and skill-building activities to promote nutrition and parenting-related behavior change. The group sessions will last between 1.5-2 hours and groups will meet biweekly for a period of 12 months. Due to the COVID pandemic, group sessions were paused for three months (March-June 2020). The intervention resumed in July 2020 with delivery via home visits rather than peer groups, and concluded in September 2020.
  Interventions: Behavioral: Nutrition+parenting, mothers
- Nutrition+parenting, mothers and fathers (Experimental): Community health workers (CHWs) will facilitate peer group sessions with mothers and fathers of children aged 0-18 months at enrollment. CHWs will deliver key messages and facilitate problem-solving and skill-building activities to promote nutrition and parenting-related behavior change. The group sessions will last between 1.5-2 hours and groups will meet biweekly for a period of 12 months. Due to the COVID pandemic, group sessions were paused for three months (March-June 2020). The intervention resumed in July 2020 with delivery via home visits rather than peer groups, and concluded in September 2020.
  Interventions: Behavioral: Nutrition+parenting, mothers and fathers
- Standard of care control (No Intervention): Local standard of care

INTERVENTIONS:
Behavioral: Nutrition, mothers — Nutrition-related social and behavior change (SBC) messages and activities for mothers focused on infant and young child feeding (IYCF), dietary diversity, water, sanitation, and hygiene (WASH), food access (use of income and home-grown foods), psychosocial well-being, gender equity, intra-household resource allocation, partner communication and household decision-making
  Arms: Nutrition, mothers
Behavioral: Nutrition, mothers and fathers — Nutrition-related social and behavior change (SBC) messages and activities for mothers and fathers focused on infant and young child feeding (IYCF), dietary diversity, water, sanitation, and hygiene (WASH), food access (use of income and home-grown foods), psychosocial well-being, gender equity, intra-household resource allocation, partner communication and household decision-making
  Arms: Nutrition, mothers and fathers
Behavioral: Nutrition+parenting, mothers — Nutrition- and parenting-related social and behavior change (SBC) messages and activities for mothers focused on infant and young child feeding (IYCF), dietary diversity, responsive caregiving and child stimulation (play and communication), water, sanitation, and hygiene (WASH), food access (use of income and home-grown foods), psychosocial well-being, gender equity, intra-household resource allocation, partner communication and household decision-making
  Arms: Nutrition+parenting, mothers
Behavioral: Nutrition+parenting, mothers and fathers — Nutrition- and parenting-related social and behavior change (SBC) messages and activities for mothers and fathers focused on infant and young child feeding (IYCF), dietary diversity, responsive caregiving and child stimulation (play and communication), water, sanitation, and hygiene (WASH), food access (use of income and home-grown foods), psychosocial well-being, gender equity, intra-household resource allocation, partner communication and household decision-making
  Arms: Nutrition+parenting, mothers and fathers

SUMMARY:
This study aims to evaluate the independent and combined effectiveness of engaging both mothers and fathers in bundled parenting and nutrition behavior change packages on early child nutrition and development.

DETAILED DESCRIPTION:
The overall aim of EFFECTS is to develop, implement, and evaluate nutrition and parenting interventions that will be delivered by community health workers in the Mara region of Tanzania. We will use a 2x2 factorial cluster randomized controlled study design, plus a local standard of care control group, to evaluate the effectiveness of EFFECTS on the primary outcomes of early child nutrition and development. In total, there will be five study arms: nutrition intervention with mothers, nutrition intervention with mothers and fathers, bundled nutrition and parenting intervention with mothers, bundled nutrition and parenting intervention with mothers and fathers, and a local standard of care control. We hypothesize that an intervention approach that engages fathers will benefit the primary outcomes; a bundled nutrition and parenting package will benefit the same primary outcomes; and that the combined intervention approach - that both engages fathers and bundles nutrition and parenting messages - will have additive benefits on the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Household has a child aged 0-18 months at study enrollment
* Child has a mother/female caregiver with a male partner
* Mother, father, and child anticipate remaining in the study area for the duration of the study
* The mother, and father where appropriate, is willing to participate in a peer group for the duration of the intervention, receiving full knowledge of the amount of time they are expected to contribute to this study.
* Both mother and father provide informed consent.
* Fathers have to be present in household with mother/child 10 months out of the year

Exclusion Criteria:

* None (only those households not meeting all the above criteria will be excluded from the study)

Ages: 0 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 960 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Change in child dietary diversity (24 hrs) | 12 months
  Child dietary diversity (24 hours) defined as the number of food groups out of eight food groups consumed in the previous day based on World Health Organization (WHO) guidelines and is assessed in children aged six months or older. A higher score reflects a higher likelihood of reaching a nutritionally adequate diet.
Change in early child development | 12 months
  Bayley Scales of Infant and Toddler Development, Third Edition is used to assess cognitive, language, and motor development. Each domain of development is reported separately. In each scale, raw scores are converted to composite scores ranging from 40-160. The average score is 100 and the standard deviation is 15. A higher score denotes higher performance.

SECONDARY OUTCOMES:
Child dietary diversity (7 days) | 12 months
  Child dietary diversity (7 days) defined as number of food groups out of a total of eight food groups consumed in the previous seven days based on WHO guidelines and is assessed in children aged six months or older. A higher score reflects a higher likelihood of reaching a nutritionally adequate diet.
Child nutrition status | 12 months
  Calculated as height-for-age Z-scores (HAZ) and weight-for-height Z-scores (WHZ), based on WHO Multicentre Child Growth Standards.
Proportion of children who meet minimum meal frequency guidelines | 12 months
  Using a caregiver self-reported questionnaire adapted from WHO-UNICEF, proportion of children aged six months or older (breastfeeding and non-breastfeeding) who meet minimum meal frequency guidelines during the previous 24 hours.
Parent-child interactions | 12 months
  Interactions of the child with each parent using the Observation of Mother-Child Interactions tool. Total scores are summed. A higher score represents better parent-child interactions.
Caregiver early childhood development (ECD) knowledge | 12 months
  Caregiver (mother and father) knowledge of early childhood development (ECD) assessed using a caregiver self-report questionnaire of the perceived expected ages at which children can attain developmental milestones. Responses within a theoretically defined age range are scored as correct, and an overall knowledge of ECD score is created by summing the total number of correct items. Higher scores represent improved knowledge of ECD.
Caregiver infant and young child feeding (IYCF) knowledge | 12 months
  Caregiver (mother and father) knowledge on two topics: 1) Breastfeeding knowledge and support score; 2) Complementary feeding knowledge score (food consistency, nutritious porridge, growth); These are based on questionnaire adapted from WHO-UNICEF. Total scores (# of correct responses) are summed; a higher score represents higher level of knowledge related to recommended IYCF practices.
Change from baseline in household food allocation of animal source foods | 12 months
  Consumption of animal source foods (ASF: eggs, meat, and fish but excluding dairy) yesterday by child given father, mother, or child consumed ASF [household ASF consumption] yesterday; Consumption of ASF yesterday by mother given household ASF consumption yesterday; Consumption of ASF yesterday by father given household ASF consumption yesterday
Responsive feeding practices | 12 months
  Responsive feeding was measured among mothers using a maternal-reported scale. Each item is scored on 4-point Likert scale: 0 = never, 1 = sometimes, 2 = often, and 3 = always. Negatively worded items were reverse scored. We created an overall responsive feeding score based on the average of 8 items, whereby higher scores indicated more responsive feeding behaviors.
Caregiver stimulation practices | 12 months
  Caregiver (mother and father) stimulation practices assessed using a caregiver self-report questionnaire of the frequency of engagement in stimulation activities (e.g., naming things, playing) with the child in the past week, adapted from the Family Care Indicators. Each item was scored on a 4-point frequency scale (0=never, 1=once or twice a week, 2=multiple times a week, and 3=every day or nearly every day) and summed for a total score. Higher scores represent more frequent engagement in stimulation.
Co-parenting | 12 months
  For the brief version of the Co-parenting Relationship Scale (CRS), each item is scored on a 4-point scale, ranging from 0=not true, 1=a little bit true, 2=mostly true, 3=very true. The items are averaged to generate a total score, which similarly ranges from 0 to 3. Higher values of the total average score indicate more positive co-parenting.
Couples' communication (frequency, quality) and decision-making | 12 months
  Couples' communication and decision-making with respect to household matters (e.g., income, food allocation) using a self-report questionnaire adapted from Promundo and asked to both mothers and fathers. Two sub-scales will be reported: (1) frequency of communication, which is the average across 8 Likert-scored items (3=often, 2=sometimes, 1=rarely, and 0=never); (2) women's decision-making power, which is the total number of decisions over which the woman had the final say independently or jointly with her partner (8 total items). Higher scores will represent more frequent couples' communication and greater women's decision-making power.
Gender equitable attitudes | 12 months
  Attitudes toward gender norms and roles assessed on both women and men. For each of the 12 items on the scale, women and men will report their level of agreement scored on a 5-point scale ranging from 1 (strongly agree) to 5 (strongly disagree). The items are summarized to generate a total score ranging from 12 to 60 or a standardized z-score. Higher values indicate more gender equitable attitudes toward gender norms and women's and men's social roles and relations within a household.
Time use patterns | 12 months
  Time use patterns using 7 day recall, particularly chores and childcare activities, using adapted version of International Food Policy Research Institute's Women's Empowerment in Agriculture (WEIA) tool, assessed on both mothers and fathers. Two main indicators of time use will be reported - time spent on work activities (which can be further grouped into domestic chores and income-generating activities) and non-work activities (leisure and rest) - which each refer to the total number of hours spent for that category of activities. Smaller differences in time spent between men and women indicate greater gender equity at household level.
Proportion of households that purify drinking water | 12 months
  Using a caregiver self-report questionnaire adapted from WHO-UNICEF, 2 items will be administered to caregivers to calculate proportion of households that purify drinking water.
Proportion of households with observed animal feces in house or compound | 12 months
  Using an observational checklist adapted from WHO-UNICEF, 1 item will assess presence of animal feces in house or compound (yes/no).
Change in frequency of caregiver handwashing with cleansing agent at critical times during the past 24 hours | 12 months
  Using a caregiver self-report questionnaire adapted from WHO-UNICEF, 3 items will be administered to measure change in frequency of handwashing with cleansing agent at critical times during the past 24 hours.
Change in frequency of child handwashing with cleansing agent at critical times during the past 24 hours | 12 months
  Using a caregiver self-report questionnaire adapted from WHO-UNICEF, 3 items will be administered to measure change in frequency of child handwashing with cleansing agent at critical times during the past 24 hours.
Caregiver water, sanitation, and hygiene (WASH) knowledge | 12 months
  Caregiver (mother and father) knowledge of recommended water, sanitation, and hygiene (WASH) practices (making food safe, avoiding sickness, washing hands). These are based on questionnaire adapted from WHO-UNICEF. Total scores (# of correct responses) are summed; a higher score represents higher level of knowledge related to recommended WASH practices.
Maternal and paternal depressive symptoms | 12 months
  Maternal and paternal depressive symptoms will be measured using the Self-Reporting Questionnaire (SRQ-20, excluding the item on suicidal ideation). The SRQ-20 comprises 20 yes/no items to assess the presence of depression and anxiety-related symptoms in the past 30 days. The 19 items used in this study will be summed to create a total score, ranging from 0 to 20.
Intimate partner violence (IPV) | 12 months
  Mothers' experience of intimate partner violence will be measured based on self-reported experiences of physical, emotional, and/or sexual violence by their male partner in the past 3 months. These questions come from IPV questionnaire in the domestic violence module of the Tanzania Demographic and Health Surveys. Maternal victimization of IPV will be analyzed according to four classifications: (1) any type of violence; (2) any physical violence; (3) any emotional violence; and (4) any sexual violence.
Parenting stress | 12 months
  The Parental Distress subscale of the Parenting Stress Index questionnaire was used with both mothers and fathers. Each item is scored on a 4-point Likert scale. Applicable items will be reverse-coded, such that the highest response option=4 is in the direction of more parenting stress and response option=1 is reflective of minimal/no parenting stress. Total scores will be calculated for the Parental Distress subscale. Higher scores indicate greater parenting stress.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Pat Kieffer, MSc., Principal Investigator — Project Concern International; Nilupa Gunaratna, PhD, Principal Investigator — Purdue University; Aisha Yousafzai, PhD, Principal Investigator — Harvard H.T. Chan School of Public Health
Locations (1):
- Project Concern International, Musoma, Mara, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeong J, Mapendo F, Hentschel E, McCann JK, Yousafzai AK. Validation of an observational tool for assessing mother-child and father-child interactions in Mara, Tanzania. Dev Psychol. 2026 Jan;62(1):221-232. doi: 10.1037/dev0001909. Epub 2025 Jan 9. PMID 39786795
- [Derived] O'Malley SF, Ambikapathi R, Ghosh S, Galvin L, Jeong J, Mosha D, PrayGod G, Mapendo F, Shively G, Murray-Kolb LE, Gunaratna NS. Contribution of Food from Market Purchases and Home Production to Child Nutrient Intake: Evidence from the EFFECTS Study Baseline Data. J Nutr. 2024 Jun;154(6):1907-1916. doi: 10.1016/j.tjnut.2024.04.015. Epub 2024 Apr 11. PMID 38608871
- [Derived] EFFECTS Study Investigators. Engaging Fathers for Effective Child Nutrition and Development in Tanzania (EFFECTS): study protocol for a five-arm, cluster-randomized trial. Trials. 2024 Mar 14;25(1):188. doi: 10.1186/s13063-022-07002-4. PMID 38486278
- [Derived] Jeong J, Ahun MN, Gunaratna NS, Ambikapathi R, Mapendo F, Galvin L, Kieffer MP, Mwanyika-Sando M, Mosha D, O'Malley SF, Verissimo CK, PrayGod G, Yousafzai AK. Effects of engaging fathers and bundling parenting and nutrition interventions on early child development and maternal and paternal parenting in Mara, Tanzania: a factorial cluster-randomized controlled trial. J Child Psychol Psychiatry. 2024 May;65(5):694-709. doi: 10.1111/jcpp.13897. Epub 2023 Oct 6. PMID 37800367
- [Derived] Galvin L, Verissimo CK, Ambikapathi R, Gunaratna NS, Rudnicka P, Sunseri A, Jeong J, O'Malley SF, Yousafzai AK, Sando MM, Mosha D, Kumalija E, Connolly H, PrayGod G, Endyke-Doran C, Kieffer MP. Effects of engaging fathers and bundling nutrition and parenting interventions on household gender equality and women's empowerment in rural Tanzania: Results from EFFECTS, a five-arm cluster-randomized controlled trial. Soc Sci Med. 2023 May;324:115869. doi: 10.1016/j.socscimed.2023.115869. Epub 2023 Mar 27. PMID 37023660
- [Derived] Ambikapathi R, Irema I, Lyatuu I, Caswell B, Mosha D, Nyamsangia S, Galvin L, Mangara A, Boncyk M, Froese SL, Verissimo CK, Itatiro J, Kariathi V, Kazonda P, Wandella M, Fawzi W, Killewo J, Mwanyika-Sando M, PrayGod G, Leyna G, Patil C, Gunaratna NS. Gender and Age Differences in Meal Structures, Food Away from Home, Chrono-Nutrition, and Nutrition Intakes among Adults and Children in Tanzania Using a Newly Developed Tablet-Based 24-Hour Recall Tool. Curr Dev Nutr. 2022 Feb 8;6(3):nzac015. doi: 10.1093/cdn/nzac015. eCollection 2022 Mar. PMID 35317413